CLINICAL TRIAL: NCT05013918
Title: Oral Health and Nutrition Integrated Care Model
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N202107030
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2021-08

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized people in Nursing Home
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention

SUMMARY:
The purpose of this project is to propose an "Oral Health and Nutrition Integrated Service Model" for the long-term care system based on the establishment of the assessment tools for oral hygiene and health, swallowing ability, nutritional status and food texture. This service model will be as the reference for long-term care policy making. This project includes four aspects such as evaluation tools, professional training, community promotion and policy development which will be completed in 5 stages. In the first stage, we will search and review the domestic and international materials which are related with the tools for evaluating oral hygiene and health (oral health assessment tool, OHAT), swallowing ability (EAT-10, eating assessment tool; functional oral intake scale, FOIS), nutritional status (Taiwan version of mini nutritional assessment, MNA) and food texture (Taiwan food texture grading system). We will also inventory the resources of oral health and nutrition before importing to community. In the second stage, an expert meeting will be held to determine the evaluation tool and the teaching materials of the training courses. In the third stage, an institution (En Chu Kong Nursing Home) will be the filed area to establish the "Oral Health and Nutrition Integrated Service Model". At the same time, assistants and instructors will be trained for conducting the assessment of oral health and nutrition status in the institution. Then, the status of oral health, chewing ability and nutrition will be investigated in the institution. In the fourth stage, we will modified the materials of training programs based on the data from resources inventory for the community (Zhong-He District, for example: Li-Xing Village, De-Xing Village or Zheng-Xing Village). Furthermore, the training programs for assistants and instructors will be also held in the community during the fourth stage. In the fifth stage, based on the evaluation tools and the integrated service models, the practical suggestions will be provided for the long-term care service policy making and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized people in En Chu Kong Nursing Home (Taiwan)
* Consciousness with expressing ability

Exclusion Criteria:

* Unconscious
* Without expressing ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized people in En Chu Kong Nursing Home (Taiwan)
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Oral hygiene and health | at enrollment
  OHAT (oral health assessment tool)
Swallowing ability | at enrollment
  EAT-10 (eating assessment tool); FOIS (functional oral intake scale)
Nutritional status | at enrollment
  MNA (mini nutritional assessment in Mandarin)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical Universty, Taipei, Taiwan

REFERENCES:
- [Derived] Chou KR, Huang MS, Chiu WC, Chen YH, Chen YY, Xiao Q, Yang SC. A comprehensive assessment of oral health, swallowing difficulty, and nutritional status in older nursing home residents. Sci Rep. 2023 Nov 14;13(1):19914. doi: 10.1038/s41598-023-47336-w. PMID 37964096